CLINICAL TRIAL: NCT05428501
Title: Awareness, Care & Treatment In Obesity Management - An Observation in Mainland China
Acronym: ACTION China
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: DAS-004; U1111-1266-4279 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-05-19; First posted 2022-06-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Person Living with Obesity (PLwO): PLwO recruited via online platforms or face-to-face channels
  Interventions: Other: no treatment given
- Health Care Professionals (HCPs): HCPs treating people who have obesity
  Interventions: Other: no treatment given

INTERVENTIONS:
Other: no treatment given — People / Person Living with Obesity (PLwO) Health Care Professionals (HCPs)

SUMMARY:
ACTION China is a cross-sectional, observational, descriptive, and exploratory survey-based study without collection of laboratory data. The study is not related to any specific treatment options or pharmaceutical product. Collection of data will be performed via quantitative online survey by a third-party vendor.

The goal of this study is to provide insights to drive awareness around the needs of People Living with Obesity (PLwO) and Health Care Professionals (HCPs) involved in obesity treatment and management.

ELIGIBILITY:
Inclusion criteria:

PLwO:

1. Informed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
2. Male or female, aged above or equal to 18 years at the time of signing informed consent
3. Lives in mainland China and is native Chinese
4. Current BMI based on self-reported height and weight of at least 28 kg/m^2 as per mainland China definition of obesity(16) (calculated using an algorithm within the survey instrument)

HCPs:

1. Informed consent obtained before any study related activities (study-related activities are any procedure related to recording/collection of data according to the protocol)
2. Male or female, aged greather than or equal to18 years at the time of signing informed consent.
3. Physician with a license to practice
4. Specialty is not surgeon (including general, bariatric or plastic surgeon)
5. Practices in mainland China with at least 5 years in clinical practice
6. Spends at least 50% of time in direct patient care (as opposed to surgical procedures, office procedures or research/administrative tasks)
7. Has seen at least 100 patients in the past month
8. Has seen at least 10 patients needing weight management (defined as a patient with a BMI greather than or equal to28 kg/m^2 with or without comorbidities) in the past month

Exclusion criteria:

PLwO

1. Previous participation in this study. Participation is defined as having given online consent in this study 2. Currently pregnant 3. Participates in intense fitness or body building programs 4. Has had significant, unintentional weight loss (due to major injury, illness, etc) in the past 6 months 5. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation HCPs

1. Previous participation in this study. Participation is defined as having given informed consent in this study.
2. Unwillingness, inability, or language barriers precluding adequate understanding or cooperation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The respondent population will include people living with obesity (PLwO) and health care professionals (HCPs) involved in obesity treatment and management
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Weight loss motivators | Day 1-day of survey
  Multi-selection from defined list
PLwO / participants who made serious weight loss effort | Day 1-day of survey
  Percentage of participants
Response to/evaluation of weight loss discussion according to predefined list of values | Day 1-day of survey
  Single selection from defined list
  1. Not at all helpful
  2. A little helpful
  3. Somewhat helpful
  4. Very helpful
  5. Extremely helpful
Effective weight loss methods | Day 1-day of survey
  Multi-selection from defined list
Obesity attitudes | Day 1-day of survey
  5-point Likert scales:
  1: Do not agree at all 5: Completely agree
Attitudes toward prescription weight loss medication and surgery | Day 1-day of survey
  5-point Likert scales:
  1: Do not agree at all 5: Completely agree
Agreement with predefined Obesity and weight management measures | Day 1-day of survey
  5-point Likert scales:
  1: Do not agree at all 5: Completely agree
Degree to which healthcare and society is meeting needs of PLwO | Day 1-day of survey
  5-point Likert scales:
  1: Not at all meeting the needs 5: Completely meeting the needs

SECONDARY OUTCOMES:
Weight loss barriers | Day 1-day of survey
  Multi-selection from defined list
Top factors for improving weight loss outcomes | Day 1-day of survey
  Multi-selection from defined list
Types of weight management goals | Day 1-day of survey
  Multi-selection from defined list
Most helpful information for participants for weight loss | Day 1-day of survey
  Multi-selection from defined list
Responsibility for improving health of PLwO (rank of individuals/organizations in order of their responsibility) | Day 1-day of survey
  Rank of multi-selection from defined list of individuals/organizations in order of their responsibility.
  Ranks 1 - 3 where "1" means most responsible and "3" means least responsible
Most helpful support for weight loss | Day 1-day of survey
  Multi-selection from defined list
Effectiveness of guidelines for treating obesity | Day 1-day of survey
  5-point Likert scales:
  1. Not at all effective
  2. A little effective
  3. Somewhat effective
  4. Very effective
  5. Extremely effective
Ways participants receive information on weight loss management | Day 1-day of survey
  Multi-selection from defined list

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Ji L, Mu Y, Chang C, Wang H, Zhao D, Liu D, Shen Z, Chen W. Perceptions, attitudes and barriers to effective obesity care among people living with obesity and healthcare professionals in China: The ACTION-China study. Diabetes Obes Metab. 2024 Oct;26(10):4694-4704. doi: 10.1111/dom.15837. Epub 2024 Aug 9. PMID 39119627
- [Derived] Luo Y, Mu Y, Chen W, Wang H, Zhao D, Liu D, Zhang J, Ji L. Attitudes towards therapeutic options for weight management, including weight loss medications and surgery, among people living with obesity and healthcare professionals in China: A secondary analysis from the ACTION-China study. Diabetes Obes Metab. 2025 Jul;27(7):3627-3634. doi: 10.1111/dom.16369. Epub 2025 Apr 15. PMID 40230237